CLINICAL TRIAL: NCT04115462
Title: A Mechanistic Study on Morphine-induced Orthogonal Neural Plasticity for Itch and Pain Processing in Humans (a Relation of Morphine-induced Itch and Pain Processing)
Brief Title: A Relation of Morphine-induced Itch and Pain Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Principal Investigator, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: N-20190049
Record Dates: First submitted 2019-09-30; First posted 2019-10-04 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Morphine; Itch
MeSH Terms: conditions — Pruritus | interventions — Morphine; Histamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morphine (Active Comparator): Each participant will receive a single dose of 20 mg morphine tablet. At estimated peak-plasma concentration testing is conducted. The subject and the assessor are both blinded to the drug administrations.
  Interventions: Drug: Morphine; Drug: Histamine; Drug: Cowhage (Mucuna Pruriens); Drug: isotonic saline
- Placebo (Placebo Comparator): Each participant will receive a single dose of an identical placebo tablet. At estimated peak-plasma concentration testing is conducted. The subject and the assessor are both blinded to the drug administrations.
  Interventions: Drug: Placebo oral tablet; Drug: Histamine; Drug: Cowhage (Mucuna Pruriens); Drug: isotonic saline

INTERVENTIONS:
Drug: Morphine — A 20 mg tablet of morphine
  Arms: Morphine
Drug: Placebo oral tablet — Matching tablet of placebo
  Arms: Placebo
Drug: Histamine — Histaminergic itch will be evoked by a 1% histamine solution. A droplet of histamine solution will be placed on the predetermined area on the forearm, and the SPT lancet will be pierced through the histamine with 120 g of pressure for 1-2 seconds.
Drug: Cowhage (Mucuna Pruriens) — 25 spicules will be inserted in the centre of the predefined skin area on the forearm. The spicules will be gently rubbed for 15-20 seconds in circular motion to facilitate epidermal penetration
Drug: isotonic saline — A droplet of saline (0.9%) as vehicle control will be placed on the predetermined area on the forearm and the lancet will be pierced through the droplet.
  Other Names: saline
Drug: Histamine — Histaminergic itch will be evoked by a 1% histamine solution. A droplet of histamine solution will be placed on the predetermined area on the mandibular area, and the SPT lancet will be pierced through the histamine with 120 g of pressure for 1-2 seconds.
Drug: Cowhage (Mucuna Pruriens) — 25 spicules will be inserted in the centre of the predefined skin area on the mandibular area. The spicules will be gently rubbed for 15-20 seconds in circular motion to facilitate epidermal penetration

SUMMARY:
In This experiment, the investigators would like to test the two following hypotheses regarding the mechanisms by which opioids cause itch:

1. Opioids cause itch by a spinal disinhibition mechanism (central nervous system (CNS) effect).
2. Opioids cause itch through a mast cell-destabilizing effect leading to release of histamine and tryptase in the skin where itch is evoked (peripheral mechanism).

DETAILED DESCRIPTION:
Intrathecal and orally administered opioids are heavily used for the treatment of several acute pain conditions. However, while opioids are effective analgesics for acute pain, they are well-known to frequently cause itch (pruritus) as a side effect according with the two hypotheses stated above. So far, these two hypotheses have never been tested in humans.The present study describes a proposed study design for the purpose of confirming these two hypotheses in parallel in human subjects.

Primary endpoints of the study:

To evaluate changes itch and pain perception, and superficial perfusion after each itch provocations.

Secondary endpoints of the study:

To evaluate the existence of a correlation between itch sensitization and analgesic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women in the age of 20-65 years
* The participants must be able to speak and understand English

Exclusion Criteria:

* Participants with any clinically significant abnormalities that in the opinion of the investigator may increase the risk associated with trial participation or may interfere with the interpretation of the trial results.
* Pregnant or lactating female persons
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous or present neurologic, musculoskeletal or mental illnesses
* Current pain and itch causing diseases or psychiatric disorders
* Participants unable to understand or follow the instructions
* Participating in another study where investigational drug is used
* Participants had known allergy/discomfort to morphine
* Lack of ability to cooperate

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Microvascular reactivity | Before and 70 minutes after morphine/placebo administration
  The evoked cutaneous inflammation (quantified by superficial blood perfusion) will be measured by full-field laser perfusion imaging.
Microvascular reactivity | 10 minutes after every itch inductions
  The evoked cutaneous inflammation (quantified by superficial blood perfusion) will be measured by full-field laser perfusion imaging.
Assessment of itch | 1 minute after every itch inductions
  Immediately following the itch provocations, participants will be instructed to rate the itch intensity for 10 minutes using a digital visual analogue scale (VAS; eVAS Software: Aalborg, University, Denmark), on a tablet. The scale will be measured from 0 to 100, where 0 represents 'no itch' and 100 'worst itch imaginable'.
Assessment of pain | 1 minute after every itch inductions
  Immediately following the itch provocations, participants will be instructed to rate the pain intensity for 10 minutes using a digital visual analogue scale (VAS; eVAS Software: Aalborg, University, Denmark), on a tablet. The scale will be measured from 0 to 100, where 0 represents 'no pain' and 100 'worst pain imaginable'.

SECONDARY OUTCOMES:
Cold (CPT) and heat (HPT) pain thesholds | 10 minutes before morphine/placebo administration
  Thermal cold and heat stimuli will be applied by a contact heat-evoked potential stimulator (PATHWAYS; Medoc Ltd, Ramat Yishai, Israel), placed 5 cm distal to the elbow on the right dorsal forearm.
Cold (CPT) and heat (HPT) pain thesholds | 60 minutes after morphine/placebo administration
  Thermal cold and heat stimuli will be applied by a contact heat-evoked potential stimulator (PATHWAYS; Medoc Ltd, Ramat Yishai, Israel), placed 5 cm distal to the elbow on the right dorsal forearm.
Pressure Pain Threshold | 10 minutes before morphine/placebo administration
  Pressure will be applied to the supinator muscle on the left forearm, 15 cm distal to the elbow by a handheld electronic pressure algometer (Somedic AB, Stockholm, Sweden) with a standard probe of 1 cm2.
Pressure Pain Threshold | 60 minutes after morphine/placebo administration
  Pressure will be applied to the supinator muscle on the left forearm, 15 cm distal to the elbow by a handheld electronic pressure algometer (Somedic AB, Stockholm, Sweden) with a standard probe of 1 cm2.

CONTACTS AND LOCATIONS:
Locations (1):
- Mech-Sense, Medicinsk Gastroenterologisk ambulatorium, Medicineshus, Aalborg Universitetshospitalet,, Aalborg, North Denmark, Denmark